CLINICAL TRIAL: NCT02823418
Title: Impact of Neuraxial Labor Analgesia on the Incidence of Postpartum Depression: a Prospective, Observational, Multicenter Cohort Study
Brief Title: Neuraxial Labor Analgesia and the Incidence of Postpartum Depression
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Collaborators: Beijing Obstetrics and Gynecology Hospital (Other); Beijing Haidian Maternal and Child Health Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Other Study IDs: 2014[712]; ChiCTR-OCH-14004888 (Registry Identifier: Chinese Clinical Trial Registry (www.chictr.org.cn))
Record Dates: First submitted 2016-06-28; First posted 2016-07-06 (Estimated); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Parturition; Analgesia, Obstetrical; Depression, Postpartum
Keywords: primipara; childbirth; neuraxial labor analgesia; postpartum depression
MeSH Terms: conditions — Agnosia; Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No neuraxial labor analgesia: For patients who do not accept neuraxial labor analgesia, analgesics will be prescribed by obstetricians according to routine practice.
  Interventions: Procedure: No neuraxial labor analgesia
- Neuraxial labor analgesia: For patients who accept neuraxial labor analgesia, epidural analgesia or combined spinal-epidural analgesia will be provided when the cervix is dilated to 1 cm or more and continued until the cervix is fully dilated to 10 cm.
  Interventions: Procedure: Neuraxial labor analgesia

INTERVENTIONS:
Procedure: No neuraxial labor analgesia — Neuraxial analgesia will not be performed. Analgesics will be prescribed by the obstetricians according to routine practice.
  Groups: No neuraxial labor analgesia
Procedure: Neuraxial labor analgesia — Epidural or combined spinal-epidural labor analgesia will be performed when the cervix is dilated to 1 cm or more and continued until the cervix is fully dilated to 10 cm.
  Groups: Neuraxial labor analgesia

SUMMARY:
Postpartum depression (PPD) affects approximately 15% of women during the first year after giving birth, and is common across cultures. The etiology of postpartum depression is not totally clear. The severe pain experienced during childbirth was reported to be associated with the development of postpartum depression. The purpose of the present study is to evaluate whether use of neuraxial labor analgesia can reduce the incidence of postpartum depression.

DETAILED DESCRIPTION:
Postpartum depression (PPD) affects approximately 15% of women during the first year after giving birth, and is common across cultures. In postpartum Chinese women, the reported incidence ranged from 6.5% to 29.5%.

The etiology of postpartum depression is not totally clear. Identified risk factors include previous maternal blues, unplanned pregnancy, lack of marital or social support, and previous psychiatric illnesses. Furthermore, the severe pain experienced during childbirth was reported to be associated with the occurrence of postpartum depression.

A recent study of the investigators found that use of epidural analgesia during labor was associated with decreased risk of postpartum depression. However, several limitations existed in that study and further evidence is needed to reconfirm the finding. The purpose of the present study is to reevaluate whether use of neuraxial labor analgesia can reduce the incidence of postpartum depression.

ELIGIBILITY:
Inclusion Criteria:

1. Primiparae between 18 and 34 years of age with term single cephalic pregnancy;
2. Admitted to the delivery room during daytime working hours (from 8 am to 5 pm).
3. Preparing to deliver vaginally.

Exclusion Criteria:

1. History of psychiatric disease (indicate those that are diagnosed before or during pregnancy by psychiatrists);
2. Presence of contraindications to epidural analgesia, which includes: (1) History of infectious disease of the central nervous system (poliomyelitis, cerebrospinal meningitis, encephalitis, etc.); (2) History of spinal or intra-spinal disease (trauma or surgery of spinal column, intra-spinal canal mass, etc.); (3) Systemic infection (sepsis); (4) Skin or soft tissue infection at the site of epidural puncture; (5) Coagulopathy.
3. Other reasons that are considered unsuitable for study participation.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Primiparae between 18 and 34 years of age with term single cephalic pregnancy who are preparing to deliver vaginally during the daytime hours.
Sampling Method: Non-Probability Sample
Enrollment: 599 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2015-05-29 (Actual); Study Completion 2017-04-25 (Actual)

PRIMARY OUTCOMES:
The incidence of postpartum depression | At 42 days after delivery
  Postpartum depression will be defined by a score of 10 or more on the Edinburgh Postnatal Depression Scale.

SECONDARY OUTCOMES:
The mode of delivery | At the time of delivery
  The mode of delivery includes spontaneous delivery, instrumental delivery, and Caesarean delivery.
Neonatal Apgar score | At 1 and 5 minutes after delivery
  The Apgar score ranges from 0 to 10, with higher score indicating a better outcome. Scores 7 and above are generally normal; 4 to 6, fairly low; and 3 and below are generally regarded as critically low and cause for immediate resuscitative efforts.
Status of baby feeding | At 24 hours and 42 days after delivery
  The mode of baby feeding include breast feeding, mixed feeding, and formula feeding.
Severity of pain | At 24 hours and 42 days after delivery
  Severity of pain is evaluated with Numeric Rating Scale (NRS), where 0 indicates no pain and 10 the most severe pain.
Persistent pain | At 42 days after delivery
  Persistence pain is defined as a NRS pain score ≥1 that persisted since childbirth.
Persistent pain affecting daily life | At 42 days after delivery
  One of the following activities (including walking, mood, sleep or concentration) is affected by persistent pain, as judged by parturients themselves.

OTHER OUTCOMES:
2-year depression | Assessed between 23 to 24 months after childbirth.
  2-year depression is assessed with the Edinburgh Postnatal Depression Scale, a score of 10 or higher is defined as the presence of depression.
Degree of social support | Assessed between 23 to 24 months after childbirth.
  Degree of social support is assessed with the Social Support Rating Scale, score range 11 to 62, with higher score indicating better social support.
Maternal body weight | Assessed between 23 to 24 months after childbirth.
  Maternal body weight
Maternal height | Assessed between 23 to 24 months after childbirth.
  Maternal height
Duration of breast-feeding | Up to 24 months after childbirth.
  Duration of breast-feeding
Start of complementary feeding | Up to 24 months after childbirth.
  Start of complementary feeding
Chronic pain after childbirth | Up to 24 months after childbirth.
  Defined as persistent or recurrent pain that lasted for more than 3 months after childbirth.
Chronic pain affecting daily life | Up to 24 months after childbirth.
  Defined as chronic pain that interfered daily life activities including walking, mood, sleep or concentration, as judged by parturients themselves.
Maternal disease after childbirth | Up to 24 months after childbirth
  Refer to any new-onset disease that occurs after childbirth and requires medical therapy or surgical procedures.
Another childbirth | Up to 24 months after the first childbirth.
  Another childbirth
Mental Development Index | Assessed between 23 to 24 months of age.
  Assessed with the Mental Scale subtest of the Bayley Scales of Infant Development-Chinese Revision. The subtest includes 163 items and assesses adaptive behavior, language and cognitive ability. The raw score of successfully completed items is converted to the standardized Mental Development Index. The average score of Mental Development Index in normal urban children is 100 with a SD of 15, with higher score indicating better development.
Psychomotor Development Index | Assessed between 23 to 24 months of age.
  Assessed with the Motor Scale subtest of the Bayley Scales of Infant Development-Chinese Revision. The subtest includes 81 items and assesses gross and fine motor skills. The raw score of successfully completed items is converted to the standardized Psychomotor Development Index. The average score of Psychomotor Development Index in normal urban children is 100 with a SD of 15, with higher score indicating better development.
Child body weight | Assessed between 23 to 24 months of age.
  Child body weight
Child height | Assessed between 23 to 24 months of age.
  Child height
Pediatric disease | Up to 24 months of age.
  Indicates any congenital or acquired disease that requires medical therapy or surgical procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD,PHD, Principal Investigator — Peking University First Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ding T, Wang DX, Qu Y, Chen Q, Zhu SN. Epidural labor analgesia is associated with a decreased risk of postpartum depression: a prospective cohort study. Anesth Analg. 2014 Aug;119(2):383-392. doi: 10.1213/ANE.0000000000000107. PMID 24797120
- [Background] Hiltunen P, Raudaskoski T, Ebeling H, Moilanen I. Does pain relief during delivery decrease the risk of postnatal depression? Acta Obstet Gynecol Scand. 2004 Mar;83(3):257-61. doi: 10.1111/j.0001-6349.2004.0302.x. PMID 14995921
- [Background] Eisenach JC, Pan PH, Smiley R, Lavand'homme P, Landau R, Houle TT. Severity of acute pain after childbirth, but not type of delivery, predicts persistent pain and postpartum depression. Pain. 2008 Nov 15;140(1):87-94. doi: 10.1016/j.pain.2008.07.011. Epub 2008 Sep 24. PMID 18818022
- [Background] Vigod SN, Villegas L, Dennis CL, Ross LE. Prevalence and risk factors for postpartum depression among women with preterm and low-birth-weight infants: a systematic review. BJOG. 2010 Apr;117(5):540-50. doi: 10.1111/j.1471-0528.2009.02493.x. Epub 2010 Jan 29. PMID 20121831
- [Background] Wong CA. Advances in labor analgesia. Int J Womens Health. 2010 Aug 9;1:139-54. doi: 10.2147/ijwh.s4553. PMID 21072284
- [Derived] Deng CM, Ding T, Liu ZH, He ST, Ma JH, Xu MJ, Wang L, Li M, Liang WL, Li XY, Ma D, Wang DX. Impact of maternal neuraxial labor analgesia exposure on offspring's neurodevelopment: A longitudinal prospective cohort study with propensity score matching. Front Public Health. 2022 Jul 29;10:831538. doi: 10.3389/fpubh.2022.831538. eCollection 2022. PMID 35968440
- [Derived] Liu ZH, He ST, Deng CM, Ding T, Xu MJ, Wang L, Li XY, Wang DX. Neuraxial labour analgesia is associated with a reduced risk of maternal depression at 2 years after childbirth: A multicentre, prospective, longitudinal study. Eur J Anaesthesiol. 2019 Oct;36(10):745-754. doi: 10.1097/EJA.0000000000001058. PMID 31356375